CLINICAL TRIAL: NCT03740971
Title: Remote Ischemic Conditioning for Acute Moderate Ischemic Stroke (RICAMIS): a Prospective, Random, Open Label, Blinded End Point, Multi-center Study
Brief Title: Remote Ischemic Conditioning for Acute Moderate Ischemic Stroke
Acronym: RICAMIS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: General Hospital of Shenyang Military Region (Other)
Responsible Party: Principal Investigator, Hui-Sheng Chen, Department director, General Hospital of Shenyang Military Region
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: k（2018）43
Record Dates: First submitted 2018-11-12; First posted 2018-11-14 (Actual); Last update posted 2021-05-05 (Actual); Status verified 2021-05

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Guideline-based therapy+RIC (Experimental): RIC is given twice a day with 200mmHg pressure.
  Interventions: Device: Remote Ischemic Conditioning treatment
- Guideline-based therapy (Active Comparator)
  Interventions: Drug: Guideline-based therapy

INTERVENTIONS:
Device: Remote Ischemic Conditioning treatment — Remote Ischemic Conditioning is given twice a day with 200mmHg pressure.
  Arms: Guideline-based therapy+RIC
Drug: Guideline-based therapy — Guideline-based therapy
  Arms: Guideline-based therapy

SUMMARY:
The current treatment based on evidence-based medicine for acute ischemic stroke mainly includes reperfusion (intravenous thrombolysis, mechanical thrombolysis), anti-platelet and stroke units. About 1/3 patients can obtain good prognosis through intravenous thrombolysis. Good prognosis can be gotten from about 50 percent of patients with big artery disease by mechanical embolization. However, only a small proportion of the population can be treated with restoration perfusion in the time window. The main purpose of antiplatelet therapy is to prevent the recurrence and progression of stroke, and stroke unit is a kind of management mode. How to improve the neurological function of patients has been a hot and difficult problem in clinical practice.

A large number of basic and clinical studies have proved that remote ischemic conditioning (RIC) has protective effect on ischemic stroke. Hahn et al showed that RIC could play a neuroprotective role in cerebral ischemia-reperfusion injury in MCAO model. Other studies have also confirmed that preconditioning RIC has a neuroprotective effect on cerebral ischemia in animal models. One open label study by Hougaard et al shows that RIC can improve the NIHSS score in acute ischemic stroke patients. One recent study found that 300 consecutive days RIC therapy for the patients with symptomatic intracranial atherosclerotic stenosis significantly reduced the recurrence rate of stroke, improved the mRS score and recovered the blood flow in the lesion site. Furthermore, several studies have also shown that RIC can not only improve the neurological function of patients with cerebral infarction after intravenous thrombolysis and mechanical thrombolysis, but also protect the secondary brain injury after carotid stenting. These results suggest that RIC has a neuroprotective effect on ischemic stroke and deserves further study.

Based on the above discussion, this study aims to explore the efficacy and safety of RIC in the treatment of acute moderate ischemic stroke.

ELIGIBILITY:
Inclusion Criteria:

1. Patient age ≥18 years;
2. From onset to treatment ≤ 48 hours;
3. Ischemic stroke confirmed by head CT or MRI;
4. 6≤NIHSS score ≤ 16;
5. Premorbid mRS ≤ 1;
6. Signed informed consent.

Exclusion Criteria:

1. Serious neurological deficits before onset ( mRS ≥ 2)；
2. The aetiology of cardiogenic embolism, such as rheumatic mitral or aortic stenosis, artificial heart valve, atrial fibrillation, atrial flutter, sick sinus syndrome, left atrial myxoma, left ventricular wall thrombus or valve neoplasm, congestive heart failure, bacterial endocarditis, etc;
3. Uncontrolled severe hypertension (Systolic pressure ≥180 mmHg or diastolic pressure ≥110 mmHg after drug treatment);
4. Subclavian artery stenosis ≥ 50% or subclavian steal syndrome;
5. Intracranial tumor, arteriovenous malformation or aneurysm;
6. Severe abnormalities in coagulation;
7. Any contraindication for remote ischemic adaptation: the upper limb has serious soft tissue injury, fracture or vascular injury, distal upper limb perivascular lesions, etc.;
8. Comorbidity with any serious diseases and life expectancy is less than half a year;
9. Participating in other clinical trials within 3 months;
10. Patients not suitable for this clinical studies considered by researcher;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1800 (Actual)
Dates: Start 2018-12-26 (Actual); Primary Completion 2021-04-19 (Actual); Study Completion 2021-04-19 (Actual)

PRIMARY OUTCOMES:
Proportion of mRS (0-1） | 90±7 days

SECONDARY OUTCOMES:
Proportion of mRS (0-2） | 90±7 days
Incidence of early neurological deterioration | 7 days
  more than 4 NIHSS score increase compared with baseline
Incidence of stroke associated pneumonia | 12±2 days
occurrence of stroke or other vascular events | 90±7 days
proportion of death of any cause | 90±7 days

CONTACTS AND LOCATIONS:
Overall Officials: Huisheng Chen, Doctor, Study Chair — Neurology Department
Locations (1):
- General Hospital of ShenYang Military Region, Shenyang, China

REFERENCES:
- [Derived] He XY, Cui Y, Wang JQ, Wang L, Chen HS. Renal Function and Efficacy of Remote Ischemic Conditioning in Acute Moderate Ischemic Stroke: A Post Hoc Analysis of RICAMIS Trial. Brain Behav. 2025 Oct;15(10):e70831. doi: 10.1002/brb3.70831. PMID 41058191
- [Derived] Zhang XW, Cui Y, Chen HS. Smoking status and the efficacy of remote ischaemic conditioning: a secondary analysis of the RICAMIS trial. Stroke Vasc Neurol. 2025 Aug 19:svn-2025-004349. doi: 10.1136/svn-2025-004349. Online ahead of print. PMID 40830061
- [Derived] Cui Y, Cui LY, Chi X, Wang Q, Zhang XW, Chen HS. Platelet-to-Neutrophil Ratio and Efficacy of Remote Ischemic Conditioning in Acute Ischemic Stroke. PLoS One. 2025 Jul 3;20(7):e0322037. doi: 10.1371/journal.pone.0322037. eCollection 2025. PMID 40608686
- [Derived] Cui Y, Wang XH, Shang ZY, Wang L, Chen HS. Baseline neurologic deficit and efficacy of remote ischemic conditioning after acute ischemic stroke: A post hoc analysis of RICAMIS. Neurotherapeutics. 2024 Jan;21(1):e00294. doi: 10.1016/j.neurot.2023.10.004. Epub 2023 Dec 19. PMID 38241163
- [Derived] Cui Y, Yuan ZM, Liu QY, Wang YJ, Chen HS. Remote Ischemic Conditioning and Outcomes in Acute Ischemic Stroke With Versus Without Large Artery Atherosclerosis. Stroke. 2023 Dec;54(12):3165-3168. doi: 10.1161/STROKEAHA.123.045040. Epub 2023 Oct 18. PMID 37850359
- [Derived] Chen HS, Cui Y, Li XQ, Wang XH, Ma YT, Zhao Y, Han J, Deng CQ, Hong M, Bao Y, Zhao LH, Yan TG, Zou RL, Wang H, Li Z, Wan LS, Zhang L, Wang LQ, Guo LY, Li MN, Wang DQ, Zhang Q, Chang DW, Zhang HL, Sun J, Meng C, Zhang ZH, Shen LY, Ma L, Wang GC, Li RH, Zhang L, Bi C, Wang LY, Wang DL; RICAMIS Investigators. Effect of Remote Ischemic Conditioning vs Usual Care on Neurologic Function in Patients With Acute Moderate Ischemic Stroke: The RICAMIS Randomized Clinical Trial. JAMA. 2022 Aug 16;328(7):627-636. doi: 10.1001/jama.2022.13123. PMID 35972485